CLINICAL TRIAL: NCT02131909
Title: PC MIROIR : Effects of Mirror Therapy in Children With Hemiplegic Cerebral Palsy
Acronym: PC MIROIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2013-A01325-40
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: unilateral cerebral palsy; children; upper-limb; mirror therapy; bimanual coordination; kinematics analysis
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mirror therapy (Experimental): 5 sessions mirror therapy 15 minutes per week for 5 weeks
  Interventions: Procedure: mirror therapy
- bimanual rehabilitation exercises (Placebo Comparator): 5 sessions control therapy 15 minutes per week for 5 weeks
  Interventions: Procedure: bimanual rehabilitation exercises

INTERVENTIONS:
Procedure: mirror therapy — During a session, the child performs a series of 10 single, bilateral and synchronous movements while viewing the reflected image
  Arms: mirror therapy
Procedure: bimanual rehabilitation exercises — During a session, the child performs a series of 10 single, bilateral and synchronous movements while watching his two hands
  Arms: bimanual rehabilitation exercises

SUMMARY:
This is a randomized and comparative prospective test, monocentric and controlled (mirror therapy versus bimanual rehabilitation exercises), in single-blind (investigator and occupational therapist " 1 " do not know the type of rehabilitation performed).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral spastic cerebral palsy as defined by SCPE (Surveillance of Cerebral Palsy in Europe)
* Aged 7 to 17 years
* MACS (Manual Ability Classification System) 1 to 3
* Extension of the wrist more than 10°
* Free, informed and written consent of the parents
* Free, informed and written consent of the child
* affiliated, via his/her parents, to the Social Security regime

Exclusion Criteria:

* Other neuromuscular disorders known
* Cognitive impairment hampering the understanding of instructions
* Upper-limb pain (EVA score >3)
* Restriction of passive range of motion
* Visual impairment not allowing the visualization of the upper limb in the mirror
* Upper-limb Botulinum toxin injection in upper limb 6 months prior to inclusion

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Measurement of the AHA (Assisting Hand Assessment) score | 5 weeks

SECONDARY OUTCOMES:
Evolution of the AHA score | baseline, 5 weeks, 10 weeks
  a variance analysis using 2 factors (time, group) is used (between the onset and 5 weeks later, between the onset and 10 weeks later)
Measurement of the maximal grasp and pinch strength | baseline, 5 weeks, 10 weeks
  with a Baseline dynamometer
Qualitative and quantitative measurement of movement | baseline, 5 weeks, 10 weeks
  by a kinematic analysis via an Optitrack system
Measurement of the manual ability | baseline, 5 weeks, 10 weeks
  by Abilhand-kids questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HR Rauscent, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

REFERENCES:
- [Result] Gaillard F, Cretual A, Cordillet S, Le Cornec C, Gonthier C, Bouvier B, Heyman R, Marleix S, Bonan I, Rauscent H. Kinematic motion abnormalities and bimanual performance in children with unilateral cerebral palsy. Dev Med Child Neurol. 2018 Aug;60(8):839-845. doi: 10.1111/dmcn.13774. Epub 2018 Apr 27. PMID 29701242